CLINICAL TRIAL: NCT02581800
Title: Effect and Experience of PreHomeCare of Preterm Infants Using Telecommunication and Smartphone Application: A Randomized Intervention Study.
Brief Title: Effect and Experience of PreHomeCare of Preterm Infants Using Telecommunication and Smartphone Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mai-Britt Hägi-Pedersen (Other)
Responsible Party: Sponsor-Investigator, Mai-Britt Hägi-Pedersen, MSN, ICU nurse, phd student, Naestved Hospital
Organization: Naestved Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PreHomeCare
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Infants, Premature; Breastfeeding; Telecommunication; Patient Discharge; Nursing
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): The control group includes hospital consultations (usual care) on the hospital 2-3 times a week (1-2 hours) and the possibility to call the neonatal ward 24 hours a day all week until the infant gets full nutrition from the breast or bottle and gains weight. The parents register nutrition on a paper between the visits to the hospital.
- App group/intervention group (Experimental): The intervention group will receive the Smartphone application at inclusion time and learn to use it in the hos-pital. When the families go home they will use the application and receive planned video consultations 2-3 times a week and the possibility to call the neonatal ward 24 hours a day all week whenever needed, until the infant gets full nutrition from the breast or bottle and gains weight. Parents will borrow a baby weight to weigh the baby at home.
  Interventions: Other: App group

INTERVENTIONS:
Other: App group
  Arms: App group/intervention group

SUMMARY:
Background: Premature infants and their patents are discharged earlier from hospital and sent home in early in-homecare programs. Research regarding the use of health IT is needed to say, whether the use of videoconference and Smartphone application is a viable option to address the parents need for support in relations to early discharge.

Aim: Test and explore early in-homecare (PreHomeCare) with videoconference and mobile application versus hospital consultations.

Method: Main study; a randomized controlled intervention study with the hypothesis; parent of premature infants who have access to electronic knowledge and participatory guidance 24-7: increases proportion of exclusive breastfeeding, Improves parent/infant interaction, enhances confidence and increases knowledge.

Sub study 1; a field study. Sub study 2; an interview study. Perspectives: It is expected that this project will be an argument in development of care for premature infants and telemedicine use in the future

DETAILED DESCRIPTION:
Effect and experience of PreHomeCare of preterm infants using telecommunication and Smartphone application: A randomized intervention study.

Premature infants and their patents are discharged earlier from hospital and sent home in early in-homecare programs.

Effect studies of early in-homecare point towards that premature infants have lower risk of infections under the period of tube feeding, higher parental satisfaction and indicate that early in-homecare of premature infants benefit of home visits with fewer readmissions and less unscheduled support, shorter length of hospital stay and longer provision of breast milk. Standard procedure in early in-homecare is home visits but in regions of Denmark with large distances to the parent/infant this is not possible. No studies have until now offered 24-7 hours home visit support. Further research regarding the use of health IT is needed to say, whether the use of videoconference (participatory guidance) and Smartphone application (knowledge and data registration) is a viable option to address the parents need for support in relations to early discharge.

Main Study: A randomized controlled intervention study. The aim is to test the effect of the use of video communication and mobile application on exclusive breastfeeding, parent/infant interaction and parental confidence with the premature infants after PreHomeCare.

Hypothesis; Compared to parents of premature infants who receive hospital consultations, the parents of premature infants who have access to electronic knowledge and participatory guidance 24-7:

1. Increases proportion of exclusive breastfeeding.
2. Improves parent/infant interaction (MABISC-mother and baby interaction scale).
3. Enhances the families' feeling of confidence in caring for their infant (KPCS - Karitane parenting confidence scale).
4. Increases parent's knowledge with regarding the premature infant and the care. Parents will be randomized to either intervention or control group via simple randomization procedure.

The intervention group will receive a mobile application and videoconference system. The application contains three parts; 1) knowledge, 2) video contact/participatory guidance and 3) data registration.

Sample Size: Applying a significance level of 5%, a two-sided two-sample proportions test revealed that a sample size of 39 in each group maintains a power of 80% to detect the difference consisting of 55% vs. 40% breastfeeding women in the two groups after 4 weeks conditional on 66% breastfeeding at discharge. This corresponds to a sample size of 65 at randomisation. To compensate for the design effect ICC(0.01) the total sample size needed is thus approximately 160 preterm infants, 80 in each group.

Inclusion criteria: Infants who fulfil criteria for early in-home care. GA > 34+0, No need for monitoring, tube feeding and started breastfeeding/bottle feeding, Danish speaking or English speaking patents (but understand the Danish text in the application).

Exclusion criteria: Infants who do not fulfil criteria for early in-home care and parents, who require extra observations of the parent-infant relationship.

Data analysis; the results of the intervention and control group will be compared and analysed following "intention to treat" principle.

Qualitative evaluation:

Sub study 1: A field observational study: The aim is describe what characterizes nursing practice in PreHomeCare from the parents' angle in home around video consultations. Method will be based on Spradley "participant observation". The focus for the observation is the nurses' communication, how is her act on the screen etc. The field observations are expected to enlighten the characteristics of the nursing practice with a systematic description of PreHomeCare setting using video consultations. The prose text will be analysed following Ricoeur.

Sub study 2: An interview study: The aim is to explore how parents of premature infants experience PreHomeCare with use of video communication and mobile application. The study will be planned and conducted with inspiration from Kvale and Brinkmann´s instructions. The main focus for the interview will be to uncover the main question: "How did you experience PreHomeCare?" with a particular focus on what have been especially meaningful for the parents under PreHomeCare. The verbatim transcribed material will be analysed following Ricoeur interpretations theory.

Perspectives: This study will access new knowledge on the effect and experience with PreHomeCare. It will give insight in what is needed to make clear goals for the quality of the treatment and care for premature infants and parents in the last part of the admission/PreHomeCare. It is expected that this project will be an argument in further development of care for premature infants and telemedicine use in the future. The increased effectiveness can address challenges and help relocate economic and professional health services.

ELIGIBILITY:
Inclusion Criteria:

* Infants who fulfil criteria for early in-home care. GA > 34+0, No need for monitoring, tube feeding and started breastfeeding/bottle feeding, Danish speaking or English speaking patients (but understand the Danish text in the application).

Exclusion Criteria:

* Infants who do not fulfil criteria for early in-home care and parents, who require extra observation of the par-ent-infant relationship.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Proportion of breastfeeding | one month after discharge

SECONDARY OUTCOMES:
Parents feeling of confidence | one month after discharge
Parent/child interaction | one month after discharge
Active knowledge concerning the premature infant | one month after discharge

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (4):
  - Herning Neonatal, Herning
  - Neonatal, Næstved
  - Neonatal, Roskilde
  - Neonatal, Viborg

REFERENCES:
- [Derived] Hagi-Pedersen MB, Dessau RB, Norlyk A, Stanchev H, Kronborg H. Comparison of video and in-hospital consultations during early in-home care for premature infants and their families: A randomised trial. J Telemed Telecare. 2022 Jan;28(1):24-36. doi: 10.1177/1357633X20913411. Epub 2020 Mar 30. PMID 32228143
- [Derived] Hagi-Pedersen MB, Norlyk A, Dessau R, Stanchev H, Kronborg H. Multicentre randomised study of the effect and experience of an early inhome programme (PreHomeCare) for preterm infants using video consultation and smartphone applications compared with inhospital consultations: protocol of the PreHomeCare study. BMJ Open. 2017 Mar 9;7(3):e013024. doi: 10.1136/bmjopen-2016-013024. PMID 28279994